CLINICAL TRIAL: NCT00489710
Title: A Phase II Study of Talabostat in Patients With Metastatic Renal Cell Carcinoma
Brief Title: Talabostat in Treating Patients With Metastatic Kidney Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: safety reasons
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0401-05-FB
Record Dates: First submitted 2007-06-20; First posted 2007-06-21 (Estimated); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Kidney Cancer
Keywords: stage IV renal cell cancer; recurrent renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — PT-100 dipeptide; Flow Cytometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Talabostat (Experimental): Talabostat 600 mcg orally, daily x 14 days (21 day cycle); 2 cycles
  Interventions: Drug: talabostat mesylate; Biological: enzyme inhibitor therapy; Diagnostic Test: flow cytometry; Diagnostic Test: laboratory biomarker analysis; Biological: non-specific immune-modulator therapy

INTERVENTIONS:
Drug: talabostat mesylate
  Other Names: Val-boroPro
Biological: enzyme inhibitor therapy
Diagnostic Test: flow cytometry
Diagnostic Test: laboratory biomarker analysis
Biological: non-specific immune-modulator therapy

SUMMARY:
RATIONALE: Talabostat may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase II trial is studying how well talabostat works in treating patients with metastatic kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the response rate in patients with metastatic renal cell carcinoma treated with talabostat mesylate.
* Determine the progression-free survival of patients treated with this drug.

Secondary

* Determine the toxicity of this drug in these patients.
* Correlate changes in specific cytokine levels and peripheral blood flow cytometry with progression-free survival.

OUTLINE: This is a nonrandomized study.

Patients receive oral talabostat mesylate once daily on days 1-14. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Blood samples are obtained from patients at baseline and after each course for biomarker correlative studies. Samples are analyzed for serum cytokines and chemokines and for T-cell subsets and natural killer (NK) cells by flow cytometry. Peripheral blood lymphocytes are obtained at baseline and after course 1 for future assessment by gene microarray analysis.

ELIGIBILITY:
Inclusion Criteria

* Pathologic diagnosis of renal cell carcinoma (clinical confirmation of metastatic disease required)
* Measurable disease, defined as ≥ 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques or ≥ 10 mm by spiral CT scan
* Progressed after ≥ 1 multikinase inhibitor regimen (i.e., sorafenib tosylate or sunitinib malate)
* No history of central nervous system or brain metastasis
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Absolute neutrophil count (ANC) ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 8.5 g/dL (no packed red blood cell transfusions within the past 4 weeks) (epoetin alfa support allowed)
* Bilirubin ≤ 1.5 times the upper limit of normal (ULN) (unless due to Gilbert's syndrome)
* aspartate aminotransferase (AST) and alanine transaminase (ALT) ≤ 3 times ULN
* Creatinine < 2.0 mg/dL
* No active serious infections
* No other malignancy within the past 5 years except basal cell or nonmetastatic squamous cell skin cancer or carcinoma in situ of the cervix
* No comorbidity or concurrent condition that would interfere with protocol assessments or procedures
* No ongoing coagulopathy
* At least 4 weeks since prior systemic therapy and recovered
* Prior radiotherapy allowed as long as the lesion treated is not used to assess response
* No prior radiotherapy to > 50% of the bone marrow
* No prior radiotherapy to index lesions unless there is clearly progressive disease within the irradiated area OR measurable disease outside the irradiated area

Exclusion Criteria

* History of CNS or brain metastasis
* Pregnant, nursing or planning on becoming pregnant
* Active serious infections
* Malignancy within the past 5 years except basal cell or nonmetastatic squamous cell skin cancer or carcinoma in situ of the cervix
* comorbidity or concurrent condition that would interfere with protocol assessments or procedures

Ages: 19 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-12 (Estimated); Primary Completion 2007-05-30 (Actual); Study Completion 2007-05-30 (Actual)

PRIMARY OUTCOMES:
Objective response rate | After 9 and 12 evaluable patients (126 to 168 days of total treatment). Each course is 14 days and repeats every 21 days in the absence of disease progression or unacceptable toxicity.
  Evaluable patients are those that have completed 4 cycles of treatment.

SECONDARY OUTCOMES:
Dose-limiting toxicity | From day 1 through 14 of each course. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Any grade 3-4 non-haematological or grade 4 haematological toxicity at least possibly related to treatment
Adverse events | From day 1 through 14 of each course. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Adverse events as assessed by NCI CTCAE v3.0

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Hauke, MD, Principal Investigator — University of Nebraska